CLINICAL TRIAL: NCT00385216
Title: Effect of Nicotine on Pain After Third Molar Extraction.
Brief Title: Nicotine as an Adjuvant Analgesic for Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAA6273
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Results first posted 2010-10-27 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dental Crowding
Keywords: Third Molar; Pain
MeSH Terms: conditions — Crowding; Pain | interventions — Nicotine; Tobacco Use Cessation Devices; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine nasal spray (Active Comparator): In one sitting the subject will receive a nicotine nasal spray, 3 mg, one application.
  Interventions: Drug: Nicotine
- Placebo spray (Placebo Comparator): In one sitting the subject will receive a placebo nasal spray (0 mg), one application.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nicotine — Nicotine nasal spray 3mg x 1 before surgery
  Other Names: Nasal spray, nicotine
  Arms: Nicotine nasal spray
Other: Placebo — Placebo nasal spray 0mg x 1 before surgery
  Other Names: Nasal spray, placebo
  Arms: Placebo spray

SUMMARY:
Third molar surgery is complicated by pain and swelling for several days after surgery. Non-steroidal antiinflammatory drugs have been useful in combination with opioids for treatment. Nicotine has antiinflammatory and pain relieving properties. We will use nicotine or placebo as a nasal spray before surgery to determine whether nicotine affects pain or inflammation.

DETAILED DESCRIPTION:
This is a randomized double blind cross-over study. In each of two sittings, the third molars on one side of the mouth are removed. In one sitting the subject will receive a nicotine nasal spray (3mg) and in the other placebo. VAS and narcotic utilization will be compared within patients.

ELIGIBILITY:
Inclusion Criteria:

* over 18
* 4 molars to be removed

Exclusion Criteria:

* pregnant
* lactating
* chronic pain
* narcotic use
* asthma
* ex-smokers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-07; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Flood, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine Nasal Spray First, Then Placebo: At the first intervention, the subject will receive a nicotine nasal spray, 3 mg, one application. At the second intervention, the subject will receive a placebo nasal spray, 0 mg, one application.
- Placebo Spray First, Then Nicotine: At the first intervention, the subject will receive a placebo nasal spray, 0 mg, one application. At the second intervention, the subject will receive a nicotine nasal spray, 3 mg, one application.
Period: First Intervention
Arm/Group | Nicotine Nasal Spray First, Then Placebo | Placebo Spray First, Then Nicotine
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Nicotine Nasal Spray First, Then Placebo | Placebo Spray First, Then Nicotine
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: The baseline characteristics for the entire study population are presented here. The nicotine and placebo study populations were identical.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Pain Reported by Patient
Description: Pain were reported on the numerical rating scale for pain (NRS) with 0=no pain and 10=worst pain.
Time Frame: Up to 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Nicotine Nasal Spray: Nicotine nasal spray (3mg) was administered as 3 sprays to each nostril before surgery in either first intervention period or second intervention period.
- Placebo: Sterile saline placebo was administered as 3 sprays to each nostril before surgery in either first intervention period or second intervention period.
Arm/Group | Nicotine Nasal Spray | Placebo
Number analyzed (Participants) | 20 | 20
score on a scale | 1.6 (0.5) | 2.9 (0.5)

2. Secondary Outcome: Heart Rate
Description: Heart rate reported in beats per minute (BPM)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Nicotine Nasal Spray | Placebo
Number analyzed (Participants) | 20 | 20
Beats per minute (BPM) | 81 (15) | 76 (15)

3. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure reported in Millimeters of Mercury (mmHg)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Nicotine Nasal Spray | Placebo
Number analyzed (Participants) | 20 | 20
Millimeters of Mercury (mmHg) | 120 (11) | 121 (12)

4. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure reported in Millimeters of Mercury (mmHg)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Nicotine Nasal Spray | Placebo
Number analyzed (Participants) | 20 | 20
Millimeters of Mercury (mmHg) | 77 (8) | 76 (10)

5. Secondary Outcome: Difference in Amount of Nausea Reported
Description: For an hour postoperatively, subjects reported information on pain and nausea, and hemodynamic variables were recorded at 15-minute intervals. Telephone follow-up was recorded for 5 days postoperatively, where patients reported information on pain, nausea, and use of hydrocodone/acetaminophen as rescue analgesia.
Time Frame: 5 days
Population: The difference in the amount of nausea was not calculated. Raw data existed during the study period of 2004 to 2009. This record was completed and published in 2010 without results for this outcome measure. The data was subsequently destroyed because the data retention period had ended. As of the current year, 2024, all the raw data for this study no longer exists. This outcome cannot be calculated without the raw data.
Arm/Group | Nicotine Nasal Spray | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Difference in Number of Hydrocodone 5 mg Acetaminophen 325 mg Tablets Taken After Surgery
Description: All patients were prescribed Hydrocodone 5 mg / Acetaminophen 325 mg and were instructed to take 1 to 2 tablets for oral pain at a maximum of every 4 to 6 hours post-surgery.
Time Frame: 5 days
Population: as for outcome 5
Groups:
- Placebo: Sterile saline nasal spray was administered as 3 sprays to each nostril before surgery in either first intervention period or second intervention period.
Arm/Group | Nicotine Nasal Spray | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 days
Arm/Group | Nicotine Nasal Spray | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes